CLINICAL TRIAL: NCT04541953
Title: TeleRehabilitation Following Arthroscopic Rotator Cuff Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20-01261
Record Dates: First submitted 2020-09-02; First posted 2020-09-09 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Rotator Cuff Injuries
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation (Active Comparator)
  Interventions: Other: Telerehabilitation Therapy
- In-Person Rehabilitation (Active Comparator)
  Interventions: Other: In-person Rehabilitation Therapy

INTERVENTIONS:
Other: Telerehabilitation Therapy — Rehabilitation services will be dispensed at patients' home utilizing video telecommunication services with real-time synchronous exchange of information - range of motion exercises and stretching.
  Arms: Telerehabilitation
Other: In-person Rehabilitation Therapy — Range of motion exercises and stretching
  Arms: In-Person Rehabilitation

SUMMARY:
Telerehabilitation is a form of tele-treatment in which rehabilitation services are dispensed at patients' home utilizing video telecommunication services with real-time synchronous exchange of information. The advantages of telerehabilitation include reducing unnecessary travel to the hospital and person to person contact while maintaining social distancing. While some of the patients are truly staying at remote areas, others are unable to manage travel in the lockdown period. Telemedicine offers the opportunity to deliver rehabilitative services in the patients' home, closing geographic, physical, and motivational gaps. Punctuality on either side is also assured since the travel times are saved on both the ends.

The purpose of the research study is to compare two standard of care rehabilitation methods (telerehabilitation vs in-person rehabilitation) following routine rotator cuff repair. Objectives include assessing range of motion and patient reported functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo Rotator Cuff repair
* Age 40-80
* Ability to comply with a standardized postoperative protocol
* Willing and able to provide consent

Exclusion Criteria:

* Pregnant patient
* Age <40 years
* Previous shoulder surgery
* Unable to speak English or perform informed consent

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Level of Range of Motion | up to 1 year post-op
  Active and passive range of motions will be tested in participants: forward flexion, abduction and internal/external rotation at 0° and 90°.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) Score | up to 1 year post-op
  VAS is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain." The total score ranges from 0-10. The higher the score, the worse the pain.
American Shoulder and Elbow Surgeons (ASES) Questionnaire Score | up to 1 year post-op
  The ASES score contains a physician-rated and patient-rated section; however, only the pain visual analog scale (VAS) and 10 functional questions will be used to tabulate the reported ASES score. The total score - 100 maximum points - is weighted 50% for pain and 50% for function. The final pain score (maximum 50 points) is calculated by subtracting the VAS from 10 and multiplying by five. For the functional portion, each of 10 separate questions is scored on an ordinal scale from 0-3 for a maximal raw functional score of 30 points. The raw score is multiplied by 5/3 to make the maximal functional score out of 50 possible points. The pain and functional portions are then summed to obtain the final ASES score. The higher the score, the worse the pain and level of function.

CONTACTS AND LOCATIONS:
Overall Officials: Kirk Campbell, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data upon reasonable request. Requests should be directed to kirk.campbell@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.